CLINICAL TRIAL: NCT04731142
Title: Type 2 Diabetes Exemplar (T2DEx): A Remote Care Service for North West London
Brief Title: Type 2 Diabetes Exemplar: A Remote Care Service for North West London
Acronym: T2DEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry); Huma (Industry); North West London Collaboration of CCGs (NWL CCGs) (Other); Imperial College Health Partners (ICHP) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20IC6484
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: An experimental feasibility study with a pre-test/post-test design using a matched control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2DEx remote care service (Experimental)
  Interventions: Device: Huma; Behavioral: Video group consultations; Behavioral: KNOW Diabetes
- Matched control group (Other): This study will create a matched control group using propensity score matching (PSM), a quasi-experimental method used to mimic the characteristics of a randomised control trial that has been shown to reduce biases. PSM uses statistical techniques to construct an artificial control group by matching each study participant with a non-treated participant of similar characteristics. PSM computes the probability that a person would enrol in a program based on pre-defined characteristics, giving a 'propensity score'.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Huma — Digital remote patient monitoring using blood pressure and blood sugar devices in combination with a smartphone app ('the Huma app'). Participants are provided with home monitoring devices and download the Huma app. Data recorded via the Huma app is self-reported and includes activity data, diet information, blood glucose measurements, blood pressure measurements, weight, and the Diabetes Distress Scale.
  Other Names: Huma app
  Arms: T2DEx remote care service
Behavioral: Video group consultations — Each patient is invited to attend a total of three VGCs during the 12-weeks lasting approximately one hour and 15 minutes each. Each session is facilitated by a Practice Nurse (PN) and consists of 6-10 people with T2DM. The self-reported Huma app (see below) and patient EPR data are used to populate a "Discussion Dashboard" which is used in each VGC to facilitate discussion. During the first VGC session, patient goals are discussed and adjusted in a group setting with topics relevant to their condition covered by the PN. Between each VGC session, patients spend time working on their goals and continuing to enter self-reported metrics into the Huma app. During the second and third VGC sessions, each patient is discussed, along with their performance against agreed goals.
  Other Names: VGC
  Arms: T2DEx remote care service
Behavioral: KNOW Diabetes — Each patient is signed up to a series of educational email campaigns to complement the VGC sessions and provide broader education around diabetes management. Patients receive two emails per week during the 12-week service on a variety of topics.
  Arms: T2DEx remote care service
Other: Standard of care — Normal primary care service provided to matched control group.
  Arms: Matched control group

SUMMARY:
The aim of T2DEx is to assess the feasibility, usability, acceptability, cost-effectiveness and safety of a digital support service for people in North West London at high risk of developing complications from Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
The Type 2 Diabetes Exemplar Programme has been designed as a collaborative effort through partners from the Discover-NOW Health Data Research Hub in North West London (NWL). The remote care service is being used in primary care to demonstrate how data and technology can improve health outcomes for people living with T2DM. The service has been designed via a cross-industry collaboration between North West London Clinical Commissioning Groups (NWL CCGs), AstraZeneca, Imperial College Health Partners and Huma. The service will be offered for patients at high risk of developing complications from T2DM (such as heart attack and stroke) and will combine video group consultations, remote monitoring via a smartphone app, and educational content such as lifestyle and diet advice.

This service seeks to strengthen population health management by providing better-tailored services and proactive interventions, particularly among population groups more at risk of the adverse impacts of COVID-19. Mortality risk from COVID-19 is approximately 25% higher in patients with T2DM and shielding has resulted in reduced primary care appointments for patients with T2DM. This has created an immediate need for primary care to adapt to provide care remotely to people with T2DM. Digital-first remote pathways could make care more accessible while finding time and cost efficiencies. By combining video group consultations and remote monitoring, we can inform the patient-clinician conversation making remote care in group settings safer, efficient and more personalised.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 with the capacity to give consent
* Patients with 'high risk' OR 'very high risk' T2DM as defined by:

  * Very high risk - T2DM with existing ASCVD OR T2DM without ASCVD but with any 3 of the following:

    * HbA1c >58
    * SBP >140
    * Non-HDL >3.35 or LDL-C >2.5
    * Nephropathy (eGFR <45, or Urine ACR >3)
    * Retinopathy
    * Neuropathy (including moderate/high risk feet, previous foot ulceration and erectile dysfunction)
    * Currently smoking
  * High risk - T2DM without ASCVD but with any 2 of the following:

    * HbA1c > 58
    * SBP >140
    * Non-HDL >3.35 or LDL-C >2.5
    * Nephropathy: eGFR <45 or Urine ACR >3
    * Retinopathy
    * Neuropathy (including moderate/high risk feet, previous foot ulceration and erectile dysfunction)
    * Currently smoking
    * Black, Asian and minority ethic (BAME) status

Exclusion Criteria:

* Participants too ill to participate in the study (i.e., presence of a life-threatening condition, expected survival less than 3 months, clinically unstable)
* Participants who have previously participated in efforts that have informed the design of this research.
* Participant without access to a smartphone.
* Non-English language (the remote monitoring technology currently does not support additional languages).
* Visual disability (the remote monitoring technology currently does not natively support visual assistance).
* Active severe mental illness (SMI).
* Alcohol / drug abuse.
* Severe frailty (identified via the Electronic Frailty Index - eFI).
* Housebound / living in nursing home.
* Currently on the REWIND Programme (a NWL total diet replacement programme for patients with type-2 diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - Hammersmith & Fulham Central Primary Care Network, London
  - Hammersmith & Fulham Partnership Primary Care Network, London
  - Harrow Collaborative Primary Care Network, London
  - Healthsense Primary Care Network, London
  - Metrocare & Celandine Health Primary Crae Network, London
  - North Connect Primary Care Network, London
  - Sphere Primary Care Network, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in June 2021 and primary completion date was 30 June 2022. Patients were recruited from 5 primary care networks (PCNs) in North West London.
Period: Overall Study
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Started | 118 | 117
Completed | 118 | 117
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T2DEx Remote Care Service | Matched Control Group | Total
Number analyzed (Participants) | 118 | 117 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 118 | 117 | 235
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 75 | 144
  Male | 49 | 42 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 118 | 117 | 235
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 118 | 117 | 235

OUTCOME MEASURES:

1. Primary Outcome: % Participants Downloading Huma App
Time Frame: 12 weeks
Population: Participants in matched control group did not have access the Huma app
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 0
Participants | 95 | 0

2. Primary Outcome: Video Group Consultation Sessions Attended
Description: the number of participants attending at least one VGC
Time Frame: 12 weeks
Population: Participants in the matched control group were not provided with VGCs
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 0
Participants | 78 | 0

3. Primary Outcome: Blood Glucose Measurements Recorded
Description: Number of participants entering at least one measurement
Time Frame: 12 weeks
Population: Patients in the matched control group did not have access to remote monitoring devices
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 0
Participants | 82 | 0

4. Primary Outcome: Blood Pressure Measurements Recorded
Description: Number of participants entering at least one blood pressure measurement
Time Frame: 12 weeks
Population: Patients in the matched control group did not have access to remote monitoring devices
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 0
Participants | 90 | 0

5. Primary Outcome: Number of Weight Measurements Recorded
Description: Number of participants entering at least one weight measurement
Time Frame: 12 weeks
Population: Patients in the matched control group did not have access to remote monitoring devices
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 0
Participants | 88 | 0

6. Primary Outcome: Number of Diabetes Distress Scale Scores Recorded
Description: Number of participants entering at least one DDS measurement
Time Frame: 12 weeks
Population: Patients in the matched control group did not have access to the Huma app to complete the DDS
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 0
Participants | 45 | 0

7. Primary Outcome: Number of Deaths
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 117
Participants | 0 | 0

8. Primary Outcome: Number of Participants With Emergency Department Admissions
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 117
Participants | 10 | 14

9. Primary Outcome: Number of Participants With Hospital Admissions
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 118 | 117
Participants | 57 | 42

10. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c from beginning to end of programme
Time Frame: 6 months
Population: HbA1c tests not taken from all participants
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 62 | 64
mg/dL | -3.7 [-7.29 to -0.09] | -1.72 [-5.15 to 1.71]

11. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol from beginning to end of programme
Time Frame: 6 months
Population: Cholesterol tests not taken from all participants
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 12 | 43
mg/dL | 0.425 [-0.056 to 0.906] | -0.0182 [-0.490 to 0.125]

12. Secondary Outcome: Change in Weight
Description: Change in weight from beginning to end of programme
Time Frame: 6 months
Population: Weight not entered by all participants
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 43 | 52
kg | -2.17 [-2.9 to -1.44] | -1.6 [-3.5 to 0.3]

13. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic BP from beginning to end of programme
Time Frame: 6 months
Population: Systolic BP tests not taken from all participants
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | T2DEx Remote Care Service | Matched Control Group
Number analyzed (Participants) | 65 | 64
mmHg | -3.35 [-7.2 to 0.49] | -4.86 [-8.97 to -0.75]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | T2DEx Remote Care Service | Matched Control Group
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/117
Other Adverse Events (participants affected / at risk) | 0/118 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT04731142/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT04731142/SAP_001.pdf